CLINICAL TRIAL: NCT05517759
Title: Implementation of a Ventilator-Associated Pneumonia Prevention Bundle Among ICU Nurses in Salmaniya Medical Complex, Bahrain: A Quasi-Experimental Study
Brief Title: Application of VAP Bundle Among ICU Nurses
Status: Completed | Type: Observational
Sponsor: University of Bahrain (Other)
Responsible Party: Principal Investigator, Zainab Mohamed Ali Alaswad, Principal Investigator, University of Bahrain
Other Study IDs: university of Bahrain
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Ventilator Associated Pneumonia
Keywords: nurses; knowledge; compliance; VAP; VAP bundle; vap prevention bundle; ICU
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Educational program — The sessions were delivered in form of face to face, group disscussion, brainstorming and smart cards. The educational package covered all aspect of knowledge regarding VAP such as definitions, risk factors m cause, manifestation, diagnostic criteria, and nursing care to prevent VAP. A PowerPoint and information pamphlet were used to display the material.

SUMMARY:
Background: Ventilator associated pneumonia (VAP) is a recognized healthcare-associated infection in lungs parenchyma that occurs in patients in which they are connected to mechanical ventilator. And this infection will occur after completing 48 hours of connection to the ventilator.

Aim study aims to evaluate the effect of implementing VAP prevention bundle training program on nurses' knowledge and compliance among nurses in intensive care unit in Salmaniya Medical complex in Bahrain.

Methodology: A quantitative quasi- experimental study was conducted in the main ICU of Salmaniya Medical complex in Bahrain. Purposive sampling technique was used, and 58 ICU staff nurses were enrolled at data collection period. Tools used for data collection was a self-administrative questionnaire to assess ICU nurses' knowledge and observational checklist was used to assess their compliance. Data were analyzed with descriptive and inferential statistics

DETAILED DESCRIPTION:
nurses were approach individually to introduce the researcher and the study objectives to them once the nurse agreed to participate in the study an informed consent was given with a contact details provided to the participants including direct researcher email and researches advisor email beside to that a special direct contact number with a what's up for the participants was given to facilitate the reach to the researcher at any time if they got any doubts. After that, compliance to the VAP bundle was evaluated to determine the current status. Participants were given a multiple-choice knowledge questionnaire to assess their knowledge and researcher was observing them during the filling period to prevent using their smart phone for searching or to avoid sharing answers between them. After that the VAP bundle implementation by nurses was observed following checklists by the researcher herself and no changes was be implanted

then the nursing stuff were educated all over the three shifts about VAP bundle throughout an educational package and the schedule of teaching session was arranged with nursing supervisor at ICU to not disturb the sequence of the work timetable. Nurses received extensive educational course in a creative way. At the early beginning of this stage a banner contains VAP bundle elements size 116cm x 160 was kept Infront of ICU's entering door, this area was chosen to the banner to attracted nurses' attentions at the beginning of the shift and to make the expectation about the education to develop in their mind. Then nurses on the specified shift were divided into two groups based on there workload one group received the lecture and the second group were with patients to avoid work disturbance then the groups were switched. Group discussion, PowerPoint presentation and brain storming questions card were given to the nurses.

then During this phase, a rollup banner size (200cm x 120 cm) contains VAP bundle elements and its benefit was kept near to the nurses station to facilitate remembrance of the elements as will as because ICU at SMC are using the classic way of documentation pens with the study logo of VAP were distributed to the participants to always keep the bundle implementation in their mind, and of course we used the pandemic situation for our benefit by providing the participants N95 and KN95 masks that have a printed logo of our study, this can increase the implementation of the bundle and their adherence if the eyes get used on the logo. As well as during this phase nurse knowledge were reassessed after the intervention by using the same questionnaire that was distributed in the pre phase. the compliance of VAP bundle was monitor by the researcher who observed and record only without interfering to avoid any potential effect on the compliance. Everyday approximately during morning, evening and night shift for several hours was spent in observing nurses performing their routine care activities.

ELIGIBILITY:
Inclusion Criteria:

* all permanent ICU nurse who assigned to mechanically ventilated patients and willing to participate in the three phases of the study

Exclusion Criteria:

* Nurse who are not willing to participate and nurses who are not willing to reach the three phases of the study and ICU nurses who been taken to serve in COVID facilities and not available in Main SMC ICU during the study

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: population was all nurses from both gender and all age with different years of experience and different Level of education. nurse are working in Salmaniya medical complex (SMC) (which is one of the main governmental hospitals in Bahrain that provide secondary and tertiary care for the citizen) and taking care of patients connected to mechanical ventilator at intensive care unit ICU
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
knowledge | 1 month
  nurses knowledge about VAP disease and their knowledge about VAP prevention bundle by using questionnaire adopted from Lan, Lai and Yang (2014) study then Knowledge was categorized as poor average and good by using knowledge cut off point (the knowledge was categorized, using Bloom's cut-off point, as good if the score was between 80 and 100%, moderate if the score was between 60 and 79%, and poor if the score was less than 60%)
compliance | 1 month
  nurses application of VAP bundle elements which are 1. Elevation of the head of the bed (30-45) degree, 2. Daily sedation vacation and assessment of weaning and extubation, 3. Usage of prophylaxis for peptic ulcer disease (PUD), 4. Usage of prophylaxis of deep vein thrombosis (DVT), 5. Oral care daily with chlorhexidine The compliance was recorded daily for each bundle element, if the bundle elements performed it recorded as "yes", whereas if it was missing it was recorded as "No", Observation checklist has been obtained from Institute for Healthcare Improvement and the name of the tool was IHI Ventilator Bundle

CONTACTS AND LOCATIONS:
Locations (1):
- Univercity of Bahrain, Manama, Southerner Governorate, Bahrain

IPD SHARING:
Plan to Share IPD: No
Once the participant completes the questionnaires, he or she was asked adherences in an envelope that was be provided by the researcher and seal the envelope, then it was be collected by the researcher only from the unite. And for further confidentiality and anonymity no participant's names was be recorded during data collection and data reporting and the consent forms with the questionnaires was separated at the time of data collection.
  The data entry to the software's SPSS was done only by the investigator herself in a password protected computer and the physical copies of the questionnaires and other tools was be stored in a locked cupboard and only the researcher and her supervisor have access to the raw data. Once the study will be published and accept to disseminate a professional journal, only the aggregated data will be presented and then the stored data will be discarded